CLINICAL TRIAL: NCT04752826
Title: Phase 1/2a Open-Label, Dose-Escalation, Multicenter, FIH, Consecutive-Cohort, Clinical Trial of BI-1808, a Monoclonal Antibody to TNFR 2 As a Single Agent and in Combination with Pembrolizumab (MK-3475-D20) in Subjects with Advanced Malignancies
Brief Title: BI-1808 As a Single Agent and with Pembrolizumab (KEYTRUDA® ) in Treatment of Advanced Malignancies(Keynote-D20)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-BI-1808-01; MK3475-D20 (Other: Merck Sharp & Dohme Corp); 2020-002090-10 (EudraCT Number)
Record Dates: First submitted 2020-12-15; First posted 2021-02-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignancies; Ovarian Cancer; T-cell Lymphoma; Melanoma
Keywords: Advanced Malignancies; T-cell Lymphoma
MeSH Terms: conditions — Ovarian Neoplasms; Lymphoma, T-Cell; Melanoma | interventions — pembrolizumab; Solutions; Injections

STUDY DESIGN:
Intervention Model Description: Phase 1/2a, dose escalation, consecutive-cohort, open-label study trial of BI-1808 as a Single Agent and in Combination with Pembrolizumab in Subjects with advanced malignancies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I, Part A - Dose escalation and safety of BI-1808 as single agent (Experimental): Dose escalation of BI-1808 administrated a single agent
  Interventions: Drug: BI-1808
- Phase I, Part B - Dose escalation and Safety of BI-1808 in combination with pembrolizumab (Experimental): Dose escalation of BI-1808 in combination with pembrolizumab.
  Interventions: Drug: BI-1808; Drug: Pembrolizumab (KEYTRUDA® ) 25 Mg/mL Solution for Injection
- Phase 2a - Part A dose expansion of BI-1808 as a single agent (Experimental): BI-1808 administered as a single agent at the hypothesized recommended phase 2 dose determined in Phase 1
  Interventions: Drug: BI-1808
- Phase 2a, Part B - Dose expansion of BI-1808 in combination with pembrolizumab (Experimental): BI-1808 administered in combination with pembrolizumab at the respective hypothesized recommended phase 2 doses determined in Phase 1
  Interventions: Drug: BI-1808; Drug: Pembrolizumab (KEYTRUDA® ) 25 Mg/mL Solution for Injection

INTERVENTIONS:
Drug: BI-1808 — BI-1808 administered as a flat-dose IV infusion once every 3 weeks
Drug: Pembrolizumab (KEYTRUDA® ) 25 Mg/mL Solution for Injection — Pembrolizumab administered as a flat-dose IV infusion once every 3 weeks.
  Arms: Phase 2a, Part B - Dose expansion of BI-1808 in combination with pembrolizumab; Phase I, Part B - Dose escalation and Safety of BI-1808 in combination with pembrolizumab

SUMMARY:
The goal of this first in human clinical trial is to test BI-1808 administered as single agent and in combination with pembrolizumab in subjects with advanced malignancies whose disease has progressed after standard therapy.

The main questions it aims to answer are:

* how safe and tolerable is BI-1808
* what is maximum tolerated or administrated dose
* to determine recommended dose for further clinical trials. Participants will receive infusions of BI-1808 alone or combination with pembrolizumab every 3 weeks.

For the purpose of this study, subjects with advanced malignancies includes subjects with advanced solid tumors and subjects with T-cell lymphoma (TCL),

DETAILED DESCRIPTION:
This is a Phase 1/2a, dose-escalation, multicenter, first-in-human, consecutive-cohort, open-label study of BI-1808, as a single agent and in combination with pembrolizumab in subjects with advanced malignancies, whose disease has progressed after standard therapy.

The study will consist of 2 phases: a Phase 1 with Parts A and B, and a Phase 2a with Parts A and B.

Phase 1 Part A consists of a dose escalation of BI-1808 as a single agent to evaluate safety and tolerability and to determine the RP2D as a single agent (sRP2D) in subjects with advanced malignancies whose disease has progressed after standard therapy.

Phase 1 Part B consists of a dose escalation of BI-1808 in combination with pembrolizumab to evaluate the safety and tolerability of the combination treatment and to allow selection of the RP2D for BI-1808 in combination with pembrolizumab (cRP2D) in subjects with advanced malignancies whose disease has progressed after standard therapy.

Phase 2a will assess BI-1808 administered as a single agent (Part A) and in combination with pembrolizumab (Part B) at the respective hypothesized RP2D(s) determined in Phase 1. Phase 2a expansion will be conducted in indication specific cohorts of subjects. The aim of the Phase 2a is to further assess the safety and tolerability of BI-1808 as a single agent (Part A) and in combination with pembrolizumab (Part B), characterize its PK and pharmacodynamics, and assess preliminary antitumor activity by ORR, DoR, and progression-free survival (PFS), as measured by RECIST v1.1 and iRECIST.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to provide written informed consent for the trial.
2. Is ≥18 years of age on the day of signing informed consent.
3. Has a histologically confirmed advanced malignancy. Subjects with CTCL [MF or SS] who satisfy the Phase 2a, Cohort 3-specific eligibility criteria may be enrolled into the Phase 1 part of the study.
4. Is intolerant of, refuses, or is not eligible for standard antineoplastic therapy.
5. Has at least 1 measurable disease lesion as defined by RECIST.
6. Is able to safely undergo a baseline tumor tissue biopsy prior to first dose of BI-1808 (on non previously irradiated lesions only). The biopsy must be performed at least 4 weeks following the last dose of tumor directed therapy.
7. Has a life expectancy of ≥12 weeks.
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
9. Has adequate organ function as confirmed by laboratory values.

Phase 2a Expansion Cohort-Specific Inclusion Criteria:

Ovarian Cancer:

Histologically confirmed and documented recurrent ovarian, fallopian tube, and peritoneal cancer.

TCL:

1. histologically confirmed diagnosis
2. Stable doses of systemic steroids (≤20 mg prednisone equivalent) and of low-to-medium potency topical steroids permitted (no change in preceding 4 weeks).
3. Stage IB-IV with failure of at least 1 systemic therapy.
4. No current large cell transformation for subjects with CTCL.
5. Prior therapy - No prior allo hematopoietic stem cell transplantation (HSCT); >90 days since auto HSCT; >4 weeks since systemic therapy and >2 weeks since skin-directed therapy.
6. Stable doses of systemic steroids (≤20 mg prednisone equivalent) and of low-to-medium potency topical steroids permitted (no change in preceding 4 weeks).
7. Previous systemic therapies include brentuximab vedotin, bexarotene, extracorporeal photopheresis (ECP), methotrexate, mogamulizumab, romidepsin, vorinostat, or systemic therapy with localized radiation treatment or skin-directed therapy.

Melanoma:

1. Histologically confirmed diagnosis of unresectable or metastatic melanoma.

   Subjects in Part A:
2. Required prior therapies will include anti-programmed death-ligand 1 (PD-1) therapy either as monotherapy or as part of a combination regimen.
3. For subjects with a known BRAF V600-activating mutation combination targeted therapy will be required in addition to anti-PD-1/programmed death-ligand 1 (PD-L1) therapy.

   Subjects in part B:
4. Subjects with prior lines of treatment are not eligible.

All Tumor Types:

Locally advanced unresectable, recurrent or metastatic immune checkpoint inhibitor-naïve solid tumors, likely to benefit from immune checkpoint inhibitor treatment, based on Investigator opinion.

b. Subjects must have received prior standard therapy appropriate for their tumor type and stage of disease, or in the opinion of the Investigator, would be unlikely to tolerate or derive clinical benefit from appropriate standard of care therapy.

c. Subjects with known activation mutations must have prior target therapy.

Exclusion Criteria:

1. Needs doses of prednisolone >10 mg daily (or equipotent doses of other corticosteroids) while on the trial other than as premedication.
2. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Has known or suspected hypersensitivity to BI-1808 or pembrolizumab
4. Has cardiac or renal amyloid light-chain amyloidosis.
5. Has received the following:

   1. Chemotherapy or small molecule products within 4 weeks of first dose of BI-1808.
   2. Radiotherapy within 2 weeks of first dose of BI-1808. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) for non-CNS disease. Subjects who have previously had radiation pneumonitis are not allowed.
   3. Immunotherapy within 4 weeks prior to the first dose of BI-1808.
6. Has not recovered from AEs to at least Grade 1 by NCI CTCAE
7. Has had Grade ≥3 autoimmune manifestations of previous immune checkpoint inhibitor treatments (eg, anti-PD-1, anti-PD-L1, or anti-CTLA-4).
8. Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
9. Has an active, known, or suspected autoimmune disease.
10. Is a female subject and has the ability to become pregnant (or already pregnant or lactating/breastfeeding). However, those female subjects who have a negative serum or urine pregnancy test before enrollment and agree to use a highly effective method of birth control for 4 weeks before entering the trial, during the trial, and for 12 months after last dose of BI-1808, are considered eligible.
11. Is a male subject with partner(s) of childbearing potential (unless he agrees to take measures not to father children by using 1 form of highly effective contraception [condom plus spermicide gel] during the trial and for 12 months after completing treatment).
12. Has had major surgery from which the subject has not yet recovered.
13. Is at high medical risk because of nonmalignant systemic disease including severe active infections on treatment with antibiotics, antifungals, or antivirals.
14. Has presence of chronic graft versus host disease.
15. Has had an allogenic tissue/solid organ transplant.
16. Has known human immunodeficiency (HIV) and/or history of hepatitis B or C infections, or has a positive test for HIV antibody, hepatitis B antigen/hepatitis B virus DNA or hepatitis C antibody or RNA.
17. Has a history of active tuberculosis (Bacillus tuberculosis).
18. Has received a live vaccine within 30 days before the first dose of study treatment.
19. Has uncontrolled or significant cardiovascular disease.
20. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the trial.
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
22. Is participating or planning to participate in another interventional clinical trial, or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study drug.
23. Has a known additional malignancy of another type, with the exception of adequately treated cone biopsied carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) and basal or squamous cell carcinoma of the skin. Male subjects with asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for >1 year prior to start of trial therapy are eligible.
24. Has a diagnosis of primary or acquired immunodeficiency disorder or taking any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
25. Has symptomatic ascites or pleural effusion, requires surgical intervention of additional medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | From the start of the study treatment for up to 2 years and 90 days.
  AEs will be assessed by the investigators by severity and will be graded according to the NCI CTCAE v5.0 or higher and causality between AEs and the exposure to the study treatment.
Identify DLTs, determine the maximum tolerated dose and select a recommended Phase 2 dose (RP2D) of BI-1808, given via intravenous (IV) infusion, as a single agent (Phase 1, Part A), and in combination with pembrolizumab (Phase 1, Part B) | Up to 104 weeks (2 years)
  Select the RP2D dose for BI-1808ing mTPI-2 design.
Occurrence of serious adverse events (SAEs) | Up to 104 weeks (2 years)
  SAEs will be assessed by the investigators by severity and will be graded according to the NCI CTCAE v5.0 or higher and causality between SAEs and the exposure to the study treatment

SECONDARY OUTCOMES:
Evaluation of PK parameters for BI-1808. Maximum observed plasma concentration (Cmax) | Up to 104 weeks (2 years)
  Study the PK profile of BI-1808 according to a non-compartmental analysis using a validated software
Evaluation of ADA response to BI-1808 in serum with validated method | Up to 104 weeks (2 years)
  The detection and characterization of antibodies to BI-1808 will be performed using a validated method and will be evaluated for BI-1808 serum concentration to enable interpretation of the antibody data
Measurement of TNFR2 receptor occupancy on CD14+ and/CD16+ cells in serum with validated method | Up to 104 weeks (2 years)
  evaluate the receptor occupancy of BI-1808 as a single agent and in combination with pembrolizumab on T-cells expressing TNFR2 in absolute value

CONTACTS AND LOCATIONS:
Overall Officials: Andres McAllister, PhD, Study Director — BioInvent International AB
Locations (19):
- United States (2):
  - City of Hope National Medical Center, Duarte, California
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
- Hungary (3):
  - PRA Health Sciences - Hungary, Budapest
  - Magyar Honvédség-Egészségügyi Központ, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
- Russia (3):
  - Byudzhetnoye Uchrezhdeniye Zdravookhraneniya Omskoy Oblasti - Klinicheskiy Onkologicheskiy Dispanser, Omsk
  - National Medical Research Center VA Almazov, Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skanes University Hospital, Lund
  - Karolinska University Hospital, Solna, Stockholm
- United Kingdom (6):
  - University Hospitals of Leicester NHS Trust, Leicester
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK, London
  - The Royal Marsden Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No